CLINICAL TRIAL: NCT02815553
Title: Cardiac Tumors Interventional （Radio Frequency/Laser Ablation）Therapy
Acronym: CTIH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Liu Liwen, MD,PhD, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20162034-1
Record Dates: First submitted 2016-05-27; First posted 2016-06-28 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Tumors
MeSH Terms: conditions — Heart Neoplasms

ARMS (1):
- Cardiac tumors (Experimental)
  Interventions: Procedure: Direct Transthoracic Cardiac Tumor Radio Frequency Ablation Therapy; Procedure: Direct Transthoracic Cardiac Tumor Laser Ablation Therapy

INTERVENTIONS:
Procedure: Direct Transthoracic Cardiac Tumor Radio Frequency Ablation Therapy
Procedure: Direct Transthoracic Cardiac Tumor Laser Ablation Therapy

SUMMARY:
Currently, surgical removal remains the main clinical treatment for cardiac tumor patients. However, part of tumors are hard to completely resect. Also, as thoracoscopic surgeries induce great operation trauma, some patients cannot tolerate or do not will to take the operation. Therefore, new methods and techniques are in urgent need.

Our center have a 12-year experience of intervention treatment for solid tumors and has conducted several animal experiments to verify the effectiveness of transthoracic puncture ablation and radiofrequency ablation for ventricular muscle.

The purpose of this study is to conduct new method of direct transthoracic cardiac tumor-targeted Radiofrequency Ablation (RFA) or Laser induced Interstitial Thermotherapy (LITT), make minimally invasive treatment plans for cardiac tumor patients, and verify the safety and validity of intervention treatment in long term.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac tumors not suitable for surgical removal
* Subject has significant clinical symptoms or obstruction (or progressive obstruction increase) in inflow or outflow tracts shown in imaging evidence
* Cardiac tumors in ventricular chambers, myocardium, or pericardium
* Subject who cannot tolerate thoracoscopic removal or volunteer for the operation
* Subject Over 12 years old

Exclusion Criteria:

* Subject who has other cardiac diseases must receive surgical removal
* Subject has end-stage heart failure
* Subject has poor physical conditions and cannot tolerate the operation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-04; Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Mortality | 24 months
Tumor size | 24 months
  If the maximum tumor size increases, the symptom gets deteriorated; If the maximum tumor size decreases, the symptom gets relieved.
Quantification of obstructive severity | 24 months
  Investigators use the peak velocity and of stenosis (by echocardiography) to quantify obstructive severity caused by the tumor. If the peak velocity increases, the symptom gets deteriorated; if the peak velocity decreases, the symptom gets relieved.

SECONDARY OUTCOMES:
Quantification of cardiac function | 24 months
  Investigators use ejection fraction(EF) to quantify the cardiac function. If EF is higher after the operation, the cardiac function gets recovered; if EF is lower after the operation,the cardiac function does't get recovered.
Quantification of tumor blood perfusion | 24 months
  Investigators use contrast-enhanced ultrasonography to quantify tumor blood perfusion. If there is no perfusion observed, the therapy is successful；if there is perfusion, the therapy is ineffective.

CONTACTS AND LOCATIONS:
Locations (1):
- Ultrasonic Diagnosis Department of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Huang J, Lei C, Hsi DH, Zheng M, Ma H, Ta S, Hu R, Han C, Li W, Li J, Qu D, Ruan F, Wang J, Wang B, Zhao X, Liu J, Zhao L, Wang Z, Yang J, Liu L. Echocardiography-Guided Radiofrequency Ablation for Cardiac Tumors. JACC CardioOncol. 2024 Apr 30;6(4):560-571. doi: 10.1016/j.jaccao.2024.03.008. eCollection 2024 Aug. PMID 39239332